CLINICAL TRIAL: NCT04829175
Title: A Long Term Prospective Observational Post Market Clinical Follow-Up (PMCF) Registry of Ethicon Gynecare Pelvic Mesh Products for The Treatment of Stress Urinary Incontinence and Pelvic Organ Prolapse
Brief Title: Ethicon Pelvic Mesh Post Market Clinical Follow-up Registry
Status: Recruiting | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ESC_2020_03
Record Dates: First submitted 2021-03-17; First posted 2021-04-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Stress Urinary Incontinence; Pelvic Organ Prolapse
Keywords: Stress Urinary Incontinence; Pelvic Organ Prolapse; SUI; POP
MeSH Terms: conditions — Urinary Incontinence, Stress; Pelvic Organ Prolapse | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Intervention — There is no intervention, beyond necessary clinical care, in this registry. The surgical procedures being performed within the registry are identical to the surgical procedures patients would receive as part of SOC.

SUMMARY:
The objective of this post market, clinical registry is to evaluate the performance of the products of the TVT family of products or vaginal vault or uterine prolapse repair (with laparotomic or laparoscopic approach including robotic assisted) using either Gynemesh PS Mesh or Artisyn Mesh in women undergoing surgery for SUI and POP.

ELIGIBILITY:
Inclusion Criteria:

Patients who satisfy all of the following criteria will be considered eligible for enrollment in this registry:

SUI

1. Stress urinary incontinence symptoms
2. Urodynamic stress incontinence confirmed with urodynamic testing
3. Female patient ≥ 21 years of age
4. Desired surgical correction of SUI using synthetic pubo-urethral vaginal sling
5. Planned surgery for primary SUI
6. Patient able and willing to participate in follow-up
7. Patient or authorized representative has signed the approved Informed consent POP

1. Uterine or vaginal vault prolapse symptoms 2. Urodynamic testing (optional) 3. Female patient ≥ 21 years of age 4. Desired surgical correction of POP using synthetic mesh 5. Planned surgery for uterine or vaginal vault prolapse with or without concomitant SUI surgery 6. Patient able and willing to participate in follow-up 7. Patient or authorized representative has signed the approved Informed consent

Exclusion Criteria

Patients meeting any of the following criteria will be considered not eligible for enrollment in this registry:

1. Physical or psychological condition which would impair registry participation or are unwilling or unable to participate in all required registry visits and are unable to complete the questionnaires
2. Any pre-operative or intra-operative findings identified by the surgeon that may preclude the use of registry products
3. History of previous synthetic, biologic or fascial sub-urethral sling (SUI) or pelvic mesh (POP)
4. Pregnancy or plans for future pregnancy
5. History of bleeding diathesis or current anti-coagulation therapy which cannot be suspended peri-operatively according to site's standard practice
6. Current genitourinary fistula or urethral diverticulum
7. Reversible cause of incontinence (i.e. drug effect) for SUI only
8. Severe vaginal atrophy
9. History of pelvic irradiation therapy
10. Contraindication to surgery

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients ≥ 21 years of age
Study Population: Female patients ≥ 21 years of age with:
  * A diagnosis of SUI, resulting from urethral hypermobility and/or intrinsic sphincter deficiency AND/OR
  * A diagnosis of vaginal vault or uterine prolapses where surgical treatment (sacrocolposuspension or sacrocolpopexy, laparotomic or laparoscopic approach including robotic assisted) is warranted AND
  * Are scheduled to have surgical treatment using an Ethicon Gynecare Pelvic Mesh Product
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2036-03-30 (Estimated); Study Completion 2036-08-30 (Estimated)

PRIMARY OUTCOMES:
Stress Urinary Incontinence(SUI)- Cough Stress Test(CST) Assessment Change | Post-surgery through registry completion, approximately 5-10 yrs
  Objective cure (success) approximately 5-10 years after surgery, defined as a negative standardized cough stress test (CST)
Pelvic Organ Prolapse (POP)- Physical Examination with Pelvic Organ Prolapse Quantification (POP-Q) Assessment Change | Post-surgery through registry completion, approximately 5-10 yrs
  Objective cure (success) approximately 5-10 years after surgery, defined as the absence of prolapse beyond the hymen as determined by a physical examination with POP-Q

SECONDARY OUTCOMES:
SUI: International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline and post-surgery through registry completion, approximately 10 yrs
SUI: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | Baseline and post-surgery through registry completion, approximately 10 yrs
SUI: Patient Global Impression of Improvement questionnaire (PGI-I) | Post-surgery through registry completion, approximately 10 yrs
SUI: Wong-Baker FACES Pain Rating Scale | Post-surgery through registry completion, approximately 10 yrs
  To assess pain on a scale from 0 (no pain) to 10 (worst pain) related to registry device or procedure
POP: Pelvic Floor Distress Inventory (PFDI-20) Questionnaire | Baseline and post-surgery through registry completion, approximately 10 yrs
POP: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) | Baseline and post-surgery through registry completion, approximately 10 yrs
POP: Patient Global Impression of Improvement questionnaire (PGI-I) | Post-surgery through registry completion, approximately 10 yrs
POP: Wong-Baker FACES Pain Rating Scale | Post-surgery through registry completion, approximately 10 yrs
  To assess pain on a scale from 0 (no pain) to 10 (worst pain) related to registry device or procedure (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Weisberg, MD, Study Director — Ethicon, Inc.
Locations (10):
- United States (4):
  - Yale University, New Haven, Connecticut
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
- Krankenhaus der barmherzigen Schwestern, Linz, Austria
- Herlev Hospital, Hillerød, Denmark
- Hopital Jeanne de Flandres, Lille, France
- Universitatsklinikum Tubingen, Tübingen, Germany
- Bio-Medical University Rome, Rome, Italy
- Karolinska Institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu